CLINICAL TRIAL: NCT03625115
Title: Reducing Disparities in Early Intervention Use: The Opening Doors to Early Intervention Study
Brief Title: The Opening Doors to Early Intervention Study
Acronym: ODEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-014807; R01MD011598 (NIH)
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Development Delay; Development, Child
Keywords: Early Intervention; Developmental outcomes; Health disparities; Early Childhood
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: The intervention will be a modified Patient Navigator model, that we will refer to as a Family Navigator (FN) model, that will engage, inform, and assist participating parents to follow-through with the process of EI referrals and services. Eligible children randomized to the intervention arm will be provided with services from a FN. The FN will maintain contact with the family, the child's primary care provider, and Early Intervention staff, if applicable, throughout the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: Research staff collecting study data will be unaware of study arm of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Control) (No Intervention): Dyads randomized into this control arm will continue with usual care consisting of information about early intervention services and routine Child Find procedures.
- Family Navigator (Intervention) (Experimental): Dyads randomized to the Intervention arm with be assigned a designated Family Navigator (FN) who will engage, inform, and assist the participating parents to follow-through with the process of EI referrals and services.
  Interventions: Behavioral: Family Navigator (FN)

INTERVENTIONS:
Behavioral: Family Navigator (FN) — The intervention will be a modified Patient Navigator model, that we will refer to as a Family Navigator (FN) model, that will engage, inform, and assist participating parents to follow-through with the process of EI referrals and services. Eligible children randomized to the intervention arm will be provided with services from a FN. The FN will maintain contact with the family, the child's primary care provider, and Early Intervention staff, if applicable, throughout the duration of the study.
  Arms: Family Navigator (Intervention)

SUMMARY:
Poor urban minority children often experience delays in their early development leading to health disparities. Publicly funded early intervention services are available to improve child development among these children in Philadelphia, but few children access and complete these services. This can be due to parents misunderstanding what the services include or may be due to difficulties parents experience in overcoming barriers to participating. This study will test the effectiveness of the Opening Doors to Early Intervention Program, a patient navigation intervention designed to improve families' engagement with early intervention services and overcome barriers to access these services, on early child development.

DETAILED DESCRIPTION:
Developmental delays are frequently encountered among young children and disproportionately affect impoverished minority children leading to disparities in early child development. To promote healthy child development, the Individuals with Disabilities Education Act (IDEA) mandated early intervention (EI) services be made available to young children with delays, but only half of at-risk children initiate and complete EI services. As a result, many at-risk children may not receive needed services to improve their development. To foster initiation and completion of EI services, Investigators developed the Opening Doors to Early Intervention Program, a patient navigation intervention based on the Health Belief Model and targeted to at-risk urban minority children. An initial pilot study among at-risk children demonstrated feasibility and generated promising results. Therefore, this Community-Based Participatory Research application proposes to test the effectiveness of this program in a single urban county using a randomized trial design. The specific aims are to 1) determine the effectiveness of the Opening Doors to early Intervention Program on child developmental status and EI referral and services use, 2) assess whether parent engagement in early intervention mediates the effects of the program, and 3) explore whether the home learning environment, parental health literacy, and poverty moderate the effects of the program. This application addresses health disparities in early childhood by testing an intervention designed to improve participation rates in EI among urban minority children and their families on measures of early child development and EI services use. Three to four primary care pediatric clinics that provide care to this diverse urban community will be recruited to participate. Three hundred sixty children who are less than 30 months of age and have been identified as developmentally at-risk and referred for EI services at participating clinics will be randomized to receive the Opening Doors to Early Intervention Program or usual care. Urban minority parents who have previously participated in EI services will be trained as patient navigators to provide education, motivation, and assistance for families with initiation and completion of EI referrals and services. Clinicians and Child Find staff will provide usual care consisting of developmental screening and referrals without assistance. Information on participant demographic characteristics, health literacy, and the home learning environment at baseline; parent engagement and EI referral and services completion at 3, 6, 9, and 12 months; and child development at 12 months will be collected during scheduled study visits. Differences in outcomes between intervention and control participants will be compared using intention-to-treat analysis. Findings from this comparative effectiveness study can be disseminated to similar large urban counties across the U.S. to inform Child Find and EI procedures and address disparities in early child development.

ELIGIBILITY:
Inclusion Criteria:

* Child is <30 months old at time of enrollment
* Child was born >35 weeks estimated gestational age
* Parent-child dyad reside in Philadelphia and present at a Children's Hospital of Philadelphia (CHOP) primary care practice located in Philadelphia
* Parents are English or Spanish speaking
* Child has recently been referred to the Philadelphia Infant Toddler Early Intervention Program in Philadelphia County

Exclusion Criteria:

* Child moves outside of Philadelphia County
* Child has received EI services in the past 2 weeks
* Child has congenital anomalies, genetic syndromes, or human immunodeficiency virus (HIV) that place them at risk of developmental delays

Max Age: 29 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 357 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Guevara, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete, cleaned, and de-identified dataset will be made available to other investigators after all analyses have been conducted and within twelve months of the end of the final year of funding to allow for publication of all study aims. To obtain this data set, other investigators will need to contact the study Principal Investigator (PI) who will provide a data sharing agreement. The data sharing agreement will permit a deidentified data set to be shared once an Institutional Review Board (IRB) protocol has been approved at the investigators' home institution and the investigators have signed a pledge to not attempt to identify individual study subjects. The data set will be made available on a Compact Disc Read-Only Memory (CD-ROM) or through a secure File Transfer Protocol (FTP) site.
Supporting Information: SAP
Time Frame: 12 months after the end of the final year of funding.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 357 parent/child dyads were enrolled in the main RCT and provided their information for data analyses.
  A dyad refers to one parent and one child who were enrolled in the study.
Pre-assignment Details: We are reporting on participant data from 357 participants, 174 in the control arm and 183 in the intervention arm.
Period: Overall Study
Arm/Group | Usual Care (Control) | Family Navigator (Intervention)
Started (number represents each parent/child dyad) | 174 (number represents each parent/child dyad) | 183 (number represents each parent/child dyad)
Completed (number represents each parent/child dyad) | 153 (number represents each parent/child dyad) | 152 (number represents each parent/child dyad)
Not Completed | 21 | 31
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Lost to Follow-up | 17 | 24

BASELINE CHARACTERISTICS:
Population: We are reporting on participant data from 357 parent/child dyads, 174 in the control arm and 183 in the intervention arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (Control) | Family Navigator (Intervention) | Total
Number analyzed (Participants) | 174 | 183 | 357
Age, Continuous [Mean (Full Range); unit: months] — age refers to the child in the parent/child dyad
  months | 20.6 [6.4 to 29.9] | 20.8 [4.8 to 29.9] | 20.7 [4.8 to 29.9]
Age, Continuous [Mean (Standard Deviation); unit: years] — age of the parent in the parent/child dyad
  years | 30.9 (6.7) | 30.9 (7.0) | 30.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants] — sex refers to the child in the parent/child dyad
  Participants
    Female | 55 | 62 | 117
    Male | 119 | 121 | 240
Sex: Female, Male [Count of Participants; unit: Participants] — sex refers to the parent of the parent/child dyad
  Participants
    Female | 162 | 172 | 334
    Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — ethnicity of the child in the parent/child dyad
  Participants
    Hispanic or Latino | 7 | 6 | 13
    Not Hispanic or Latino | 167 | 177 | 344
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — ethnicity of the parent in the parent/child dyad
  Participants
    Hispanic or Latino | 16 | 16 | 32
    Not Hispanic or Latino | 158 | 166 | 324
    Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — race of the child in the parent/child dyad
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 7 | 6 | 13
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 107 | 132 | 239
    White | 34 | 27 | 61
    More than one race | 26 | 18 | 44
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — race of the parent in the parent/child dyad
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 8 | 7 | 15
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 111 | 136 | 247
    White | 37 | 28 | 65
    More than one race | 14 | 5 | 19
    Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Number; unit: participants] — refers to region of enrollment for the parent/child dyad
  participants
    United States | 174 | 183 | 357
Caregiver Education Level [Count of Participants; unit: Participants] — education level of the parent in the parent/child dyad
  Participants
    Less than high school | 16 | 5 | 21
    High school and/or some college | 110 | 132 | 242
    College or graduate degree | 48 | 46 | 94
Caregiver income [Count of Participants; unit: Participants] — income of the parent in the parent/child dyad
  Participants
    $14,999 or less | 36 | 32 | 68
    $15,000 - $34,999 | 58 | 68 | 126
    $35,000 - 54,999 | 40 | 37 | 77
    $55,000 or more | 37 | 45 | 82
    information not provided | 3 | 1 | 4
Caregiver Marital Status [Count of Participants; unit: Participants] — marital status of the parent in the parent/child dyad
  Participants
    Single | 79 | 97 | 176
    Separated or Divorced | 5 | 5 | 10
    Living Together As if Married or Married | 90 | 81 | 171

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Child's Cognitive Functioning (i.e., Sensorimotor Development, Problem Solving Skills)
Description: The Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) is a validated assessment of infant and toddler development for use with 1-42 month olds. The Cognitive domain consists of developmental play tasks that are administered to obtain a developmental quotient in order to determine the child's level of cognitive functioning. The composite score of the Cognitive domain is derived from a single scaled test score from the Cognitive Scale (as opposed to being comprised of the summation of scaled scores from multiple subscales, such as with the BSID-III Language and Motor composite scores). The total composite score may range from 40 to 160. Higher values denote stronger skills and abilities in the domain, indicating better outcomes. Composite scores are scaled to a mean of 100 and a standard deviation of 15.
Time Frame: 12 months
Population: A total of 223 participants completed the cognitive section of the Bayley III assessment. The reason why this number is not equal to 357 is because some families were unable to make it in person for the assessment or the assessment could not have been completed due to child behavior.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Usual Care (Control) | Family Navigator (Intervention)
Number analyzed (Participants) | 107 | 116
score on a scale | 83.50 [55 to 115] | 81.94 [55 to 110]
Statistical Analysis 1: Comparison: Usual Care (Control) vs Family Navigator (Intervention); Test type: Equivalence — A two-tailed t-test was done to compare the mean Bayley cognitive scores between the groups; p = 0.30, t-test, 2 sided

2. Primary Outcome: Early Intervention Referral Completion
Description: Completion of early intervention referrals defined as completing a multidisciplinary assessment (MDE).
Time Frame: up to 12 months
Population: We were only able to collect data from 347 participants. The reason this number does not equal 357 participants is due to participants dropping out or being withdrawn from the study before we collected early intervention data from their provider's entities.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Control) | Family Navigator (Intervention)
Number analyzed (Participants) | 170 | 177
Participants
  MDE Completed | 114 | 143
  MDE Not Completed | 56 | 34
Statistical Analysis 1: Comparison: Usual Care (Control) vs Family Navigator (Intervention); Chi-square test of independence to determine if there was a significant difference between intervention arms for those who completed a multidisciplinary evaluation (referral completed); Test type: Superiority; p = .004, Chi-squared; Pearson chi square (1) = 8.51

3. Primary Outcome: Early Intervention Services Initiation
Description: Initiation of early intervention services if deemed eligible for services, defined as participants who started services.
Time Frame: up to 12 months
Population: 207 participants were analyzed; this number came from the 207 participants who had completed their EI referral AND had been eligible for EI services or regular tracking. 200 for eligible for early intervention services and 7 were eligible for developmental tracking every 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Control) | Family Navigator (Intervention)
Number analyzed (Participants) | 93 | 114
Participants
  Started EI Services | 88 | 107
  Did not Start EI Services | 5 | 7
Statistical Analysis 1: Comparison: Usual Care (Control) vs Family Navigator (Intervention); Chi-square test of independence to determine if there was a significant difference between intervention arms for those who began early intervention services; Test type: Superiority; p = .82, Chi-squared; Pearson chi square (1) = .05

4. Primary Outcome: Evaluation of the Child's Overall Language Functioning (Receptive and Expressive Language Skills and Abilities)
Description: The BSID-III language scale will be used to assess both the understanding of language (receptive language) and use or expression of language (expressive language) skills, such as following simple directions, and naming or identifying objects and pictures. The total composite score of the Language functioning domain is composed of the sum of both the Receptive Language and the Expressive Language subscales' scaled scores. The total Language composite score may range from 40 to 160. Higher values denote stronger skills and abilities in the domain, indicating better outcomes. Composite scores are scaled to a mean of 100 and a standard deviation of 15.
Time Frame: 12 months
Population: A total of 220 participants completed the language section of the Bayley III assessment. The reason why this number is not equal to 357 is because some families were unable to make it in person for the assessment or the assessment could not have been completed due to child behavior.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Usual Care (Control) | Family Navigator (Intervention)
Number analyzed (Participants) | 107 | 113
score on a scale | 79.39 [47 to 118] | 78.71 [47 to 132]
Statistical Analysis 1: Comparison: Usual Care (Control) vs Family Navigator (Intervention); Test type: Equivalence — A two-tailed t-test was done to compare the mean Bayley language scores between the groups; p = 0.69, t-test, 2 sided

5. Secondary Outcome: Public Policy Changes
Description: Changes in state policy regarding early intervention services. During the time of the study, the COVID-19 pandemic began, which affected early intervention services and policies. This timeline is broken down into the following time periods.
  Period 1-Early Intervention in person pre pandemic: Study start date - March 19th, 2020 Period 2-Early Intervention complete closure: March 20th, 2020 - early April 2020 Period 3: Early Intervention Virtual Only: early April 2020 - June 2nd, 2020 Period 4: Early Intervention Hybrid: June 3rd, 2020 - current (in line with Governor Wolf's process to reopen plan, this was when services and evaluations were done both virtually and in person)
Time Frame: up to 12 months
Population: This analysis includes participants who were randomized into a study condition. Three participants were withdrawn immediately after enrollment, leaving a total of 357 participants randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Control) | Family Navigator (Intervention)
Number analyzed (Participants) | 174 | 183
Participants
  Participants enrolled during Period 1 | 60 | 65
  Participants enrolled during Period 2 | 0 | 0
  Participants enrolled during Period 3 | 0 | 0
  Participants enrolled during Period 4 | 114 | 118

6. Other Pre Specified Outcome: An Evaluation of Parent/Family Engagement in the Early Intervention Process
Description: Scale Name: Parent Early Intervention (EI) Engagement Questionnaire Description: Modified and validated version of the Client Engagement in Child Protective Services (CECPS) questionnaire which evaluates the caregiver(s) perceived extent of involvement, in the early intervention process.
  Scale Ranges: 9 items, split up in to 3 factors/categories, are scored on a likert scale from 1-5. Two items are reverse scored during analysis. 1 indicates poor engagement (poor outcome) and 5 indicates high engagement (high outcome).
  Each item can be scored 1-5. When items are analyzed by factor/category, the average is taken from all items in that factor/category (can be anywhere in the range of 1-5).
Time Frame: up to 3 months
Population: This data came from participants who had completed the parent engagement questionnaire at the 3 month follow up timepoints. Not all participants completed this survey, which is why the total number of participants analyzed is 333 and not 357.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (Control) | Family Navigator (Intervention)
Number analyzed (Participants) | 168 | 165
score on a scale
  Factor 1 | 4.16 (1.01) | 4.18 (1.07)
  Factor 2 | 4.68 (.77) | 4.68 (.85)
  Factor 3 | 3.74 (1.09) | 3.98 (1.11)
Statistical Analysis 1: Comparison: Usual Care (Control) vs Family Navigator (Intervention); Analysis of factor 1 items from the parent engagement questionnaire. Factor 1 (Buy-in) I am open to getting EI for my child. EI can help my child. EI can teach me new ways to help my child; Test type: Equivalence — two tailed t-test to compare the means of factor 1 between groups; p = .858, t-test, 2 sided
Statistical Analysis 2: Comparison: Usual Care (Control) vs Family Navigator (Intervention); Analysis of factor 2 items from the parent engagement questionnaire. Factor 2 (early intervention consequences): EI could have negative consequences for my child. Getting EI for my child reflects negatively on me as a parent; Test type: Equivalence — two tailed t-test to compare the means of factor 2 between groups; p = .995, t-test, 2 sided
Statistical Analysis 3: Comparison: Usual Care (Control) vs Family Navigator (Intervention); Analysis of factor 3 items from the parent engagement questionnaire. Factor 3 (Knowledge/Self-Efficacy): I know how to get EI for my child. I understand how the EI process works. If I have questions about EI, I know who to call. 12. I know my child's rights to EI under the law; Test type: Equivalence — two tailed t-test to compare the means of factor 3 between groups; p = .049, t-test, 2 sided

7. Other Pre Specified Outcome: Measure of Adversity Experienced in Childhood
Description: Scale Name: Adverse Childhood Experiences (ACEs) Scale Ranges: 0-19, average total score is reported Higher values indicate more risk (worse outcome) and lower values indicate less risk (better out ones).
Time Frame: up to 12 months
Population: 312 families completed the ACES survey. Some families did not complete this self-report measure, which is why this number is less than 357.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Usual Care (Control) | Family Navigator (Intervention)
Number analyzed (Participants) | 156 | 156
score on a scale | 4.44 [0 to 19] | 4.11 [0 to 19]
Statistical Analysis 1: Comparison: Usual Care (Control) vs Family Navigator (Intervention); A logistic regression was run to determine if the intervention arm, adjusted for child sex, income, maternal education, and primary care site, was associated with the completion of early intervention referrals for families with an adverse childhood experience survey score of greater than 2; Test type: Superiority; p = .02, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.09 to 3.21]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 12 months.
Arm/Group | Usual Care (Control) | Family Navigator (Intervention)
All-Cause Mortality (participants affected / at risk) | 0/174 | 0/183
Serious Adverse Events (participants affected / at risk) | 0/174 | 0/183
Other Adverse Events (participants affected / at risk) | 0/174 | 0/183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT03625115/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT03625115/SAP_001.pdf
  • Informed Consent Form (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT03625115/ICF_002.pdf